CLINICAL TRIAL: NCT06084559
Title: Effect of Supplemental Oxygen Therapy (SOT) in Patients With Pulmonary Vascular Diseases (PVD) Defined as Pulmonary Arterial Hypertension or Chronic Thromboembolic Pulmonary Hypertension (PH) Who Permanently Live >2500m on Pulmonary Artery Pressure (PAP) and Other Hemodynamics by Echocardiography
Brief Title: HA Residents With PVD, Pulmonary Artery Pressure (PAP) Assessed at HA (2840m) With and Without Supplemental Oxygen Therapy (SOT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PVD_HA_SOT_PAP
Record Dates: First submitted 2023-08-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Vascular Disorder; Pulmonary Artery Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: pulmonary hypertension; hypoxia; supplemental oxygen; 6-minute walk distance
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Hypoxia | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Each participant works as its own perfect control
Who Masked: Participant
Masking Description: Sham SOT (placebo, ambient hypoxic air at 2840m) versus high-flow oxygen 10l/min both via a facial mask with reservoir will be applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (ambient hypoxic air at 2840m) (Sham Comparator): Ambient hypoxic air at 2840 m will be applied via a facial mask with reservoir
  Interventions: Other: Sham Oxygen therapy
- SOT (high flow supplemental oxygen therapy) (Experimental): SOT (supplemental oxygen therapy) at a flow of 10 l/min will be applied via a facial mask with reservoir
  Interventions: Other: Supplemental oxygen therapy

INTERVENTIONS:
Other: Supplemental oxygen therapy — Mobile oxygen via pressurized bottle or mobile oxygen concentrator will be applied
  Arms: SOT (high flow supplemental oxygen therapy)
Other: Sham Oxygen therapy — Patients will reveice pressurized air via a nasal cannula
  Other Names: Placebo
  Arms: Placebo (ambient hypoxic air at 2840m)

SUMMARY:
To study the effect of SOT in patients with pulmonary vascular diseases (PVD) defined as pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension (PH) who permanently live >2500m on pulmonary artery pressure (PAP) and other hemodynamics by echocardiography and in relation to blood gases at 2840m with and without SOT.

DETAILED DESCRIPTION:
Patients with PVD diagnosed with precapillary PH with right heart catheterization and classified to groups 1 and 4 (PAH or CTEPH) who permanently live at HA >2500 (PVDHA) will have echocardiografy to assess PAP, cardiac output and other hemodynamics and arterial blood gas to assess SaO2, PaO2 and PaCO2 near their living altitude in Quito at 2840m whilst breathing ambient air or SOT at 10l/min flow via a face mask with reservoir.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-80 years old of both genders,
* Residence > 2500m of altitude
* diagnosed with precapillary PH (mean pulmonary artery pressure (mPAP) >20 mmHg, pulmonary artery wedge pressure (PAWP) ≤15 mmHg and pulmonary vascular resistance (PVR) ≥2 wood units (WU) by right heart catheterization) with PH being classified as PAH or CTEPH according to guidelines
* Patients stable on therapy
* New York Heart Association (NYHA) functional class I-III
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* Age <18 years or >80 years
* unstable condition
* Patients who cannot follow the study investigations, patient permanently living < 2500m.
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, severe smokers (>20 cigarettes/day)
* Severely hypoxemic patients at Quito permanently have persistent oxygen saturation by pulseoximetry (SpO2) <80% on ambient air.
* Patients with chronic mountain sickness (Hemoglobin > 19 g/dl in women, >21 g/dl in men)
* Patient with a non-corrected ventricular septum defect
* Relevant concomitant other disease of the heart, kidney, liver, blood (anemia hemoglobin<11 g/dl)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary Artery Pressure with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Change in PAP in mmHg assessed by echocardiography with SOT compared to ambient air (placebo) 10l/min via facial mask

SECONDARY OUTCOMES:
Change in Cardiac Output with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Change in cardiac output (l/min) assessed by echocardiography with SOT compared to ambient air (placebo) 10l/min via facial mask
Change in right to left heart diameter ratio with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Change in right to left heart diameter ratio assessed by echocardiography with SOT compared to ambient air (placebo) 10l/min via facial mask
Change in tricuspid annular plane systolic excursion (TAPSE) with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Change in tricuspid annular plane systolic excursion (TAPSE) with SOT compared to ambient air (placebo) 10l/min via facial mask
Change in right atrial area with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Change in right atrial area by echocardiography with SOT compared to ambient air (placebo) 10l/min via facial mask
Change in right heart strain with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Change in in right heart strain by echocardiography with SOT compared to ambient air (placebo) 10l/min via facial mask
Change in ph by arterial blood gases with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Changes in ph by arterial blood gases SaO2, PaO2, PaCO2 with SOT compared to ambient air (placebo) 10l/min via facial mask
Change in PaO2 by arterial blood gases with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Changes in PaO2 by arterial blood gases with SOT compared to ambient air (placebo) 10l/min via facial mask
Change in PaCO2 by arterial blood gases with SOT vs. placebo | at 15 min of breathing ambient air or supplemental oxygen
  Changes in PaCO2 by arterial blood gases with SOT compared to ambient air (placebo) 10l/min via facial mask

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Departement of Pulmonology; Rodrigo Hoyos, Dr., Principal Investigator — Carlos Adrade Marin Hospital of Quito, Equador
Locations (1):
- University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon request and based on a clear intention reviewed by an ethical review board.
  Otherwise, we will share anonymized research data after publication on a open access repository according to FAIR principles.
  Decision about the best suitable plattform is ongoing.

REFERENCES:
- [Derived] Muller J, Lichtblau M, Saxer S, Schmucki M, Furian M, Schneider SR, Herzig JJ, Bauer M, Saragoni D, Schwarz EI, Cajamarca E, Hoyos R, Ulrich S. The acute effect of high-dose supplemental oxygen on haemodynamics assessed by echocardiography in patients with pulmonary vascular disease living in Quito at 2850 m: a randomized, single-blind, placebo-controlled crossover trial. Eur Heart J Open. 2024 Dec 2;4(6):oeae097. doi: 10.1093/ehjopen/oeae097. eCollection 2024 Nov. PMID 39698150